CLINICAL TRIAL: NCT04110782
Title: Evaluation of Previeus Radical Prostatectomy and/or External Beam Radiotherapy as Protective Factors in mCRPC Patients Treated With 223Radium-dicloride and Correlation With Overall Survival: an Italian Multicenter Study
Brief Title: Radical Prostatectomy and External Beam Radiotherapy in mCRPC With 223Radium-dicloride (RaProRad)
Acronym: RaProRad
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Collaborators: University of Bari Aldo Moro (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other); University of Bologna (Other); Università degli Studi di Sassari (Other); Ospedale Civile Spirito Santo (Other)
Responsible Party: Principal Investigator, De Vincentis Giuseppe, Associate Professor, Azienda Policlinico Umberto I
Other Study IDs: MP2018SAP
Record Dates: First submitted 2019-06-20; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: 223-Radium-dicloride; Radical prostatectomy; overall survival
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium223
  Interventions: Other: Radium223

INTERVENTIONS:
Other: Radium223 — 55 kBq/ Kg

SUMMARY:
The investigators provided a multicenter analysis aiming to investigate, in a clinical practice setting, the prognostic relevance of previous primary radical prostatectomy (RP) or external beam radiotherapy (RT) in terms of Overall Survival as opposed to patients with no primary treatment performed, in a cohort of patients enrolled in 223-Ra treatment for mCRPC. 223-Ra has been administered from investigators according to the current label authorization and all patients underwent 223-Ra treatment, until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmation of prostatic adenocarcinoma, at least two symptomatic bone secondary lesions detected by bone scan and no known visceral metastases, except for malignant lymphadenopathy with less than 3 cm in the short axis diameter

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score >2 and inadequate hematological, hepatic and renal function

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Prostate cancer
Study Population: mCRPC patients admitt to Radium223 Therapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of overal survivall | From date of first 223Ra administration until the date of death from any cause or the date of the first documented progression disease, assessed up to 48 months
  The survival function, possibly stratified by categorical covariates of interest, was computed using the Kaplan-Meier product-limit estimator.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Vincentis, MD, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Clinical and anagraphical data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 12 months after publication

REFERENCES:
- [Background] Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, Bottomley D, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Coleman R, Vogelzang NJ, O'Bryan-Tear CG, Staudacher K, Garcia-Vargas J, Shan M, Bruland OS, Sartor O; ALSYMPCA Investigators. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013 Jul 18;369(3):213-23. doi: 10.1056/NEJMoa1213755. PMID 23863050
- [Background] Parker CC, Coleman RE, Sartor O, Vogelzang NJ, Bottomley D, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Bruland OS, Petrenciuc O, Staudacher K, Li R, Nilsson S. Three-year Safety of Radium-223 Dichloride in Patients with Castration-resistant Prostate Cancer and Symptomatic Bone Metastases from Phase 3 Randomized Alpharadin in Symptomatic Prostate Cancer Trial. Eur Urol. 2018 Mar;73(3):427-435. doi: 10.1016/j.eururo.2017.06.021. Epub 2017 Jul 11. PMID 28705540